CLINICAL TRIAL: NCT00617591
Title: Phase II Study of Pegylated Liposomal Doxorubicin (Doxil®), Low Frequency Dexamethasone and Revlimid® (Dd-R) in Newly Diagnosed Multiple Myeloma
Brief Title: Pegylated Liposomal Doxorubicin, Low Freq Dexamethasone & Revlimid (Dd-R) in Newly Diagnosed Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene Corporation (Industry); Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14986; 106095d (Other: USF IRB); RV-MM-PI-107 (Other: Celgene Corp.); 07OBCA990185 (Other: Ortho Biotech, Inc.)
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Myeloma
Keywords: Lenalidomide; Revlimid; Pegylated Liposomal Doxorubicin; Doxil; Dexamethasone; Decadron
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; liposomal doxorubicin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction and Maintenance Therapy (Experimental): Induction Phase Followed by Maintenance Therapy.
  Patients received lenalidomide 25 mg orally on days 1-21, dexamethasone 40 mg orally on days on 1-4, and Pegylated Liposomal Doxorubicin (PLD) 40 mg/m^2 intravenously on day 1 (reduced to 30 mg/m^2 after the initial 29 patients were treated). Cycles were repeated every 28 days.
  At the best response (4-8 cycles of induction), patients could proceed with either high-dose therapy or maintenance with lenalidomide and dexamethasone at the tolerated doses on the same schedule until disease progression.
  Dd-R: Lenalidomide (Revlimid®) combined with Pegylated Liposomal Doxorubicin (Doxil®) and Dexamethasone (Decadron®) as outlined in the Detailed Description.
  Interventions: Drug: Lenalidomide; Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — 25 mg orally on days 1-21
  Other Names: Revlimid®
Drug: Pegylated Liposomal Doxorubicin (PLD) — 40 mg/m^2 intravenously on day 1 (reduced to 30 mg/m^2 after the initial 29 patients were treated)
  Other Names: Doxil®
Drug: Dexamethasone — 40 mg orally on days on 1-4
  Other Names: Decadron®

SUMMARY:
The purpose of the research study is to determine the response rates when Revlimid® is combined with Doxil® and Dexamethasone (Dd-R) in newly diagnosed Multiple Myeloma. The study will also evaluate the side effects caused by the combination of these three drugs. This therapy is investigational in the treatment of Multiple Myeloma.

Revlimid® is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Revlimid® is approved by the Food and Drug Administration (FDA) for specific types of myelodysplastic syndrome (MDS) and Multiple Myeloma, two different types of blood cancer. It is currently being tested in a variety of other cancer conditions. In this case it is considered experimental.

Doxil® is a form of chemotherapy. It is approved by the FDA for the treatment of relapsed/ refractory Multiple Myeloma in combination with Velcade.

Dexamethasone is a steroid. It is also approved by the FDA, but not for the treatment of Multiple Myeloma. It is considered a standard part of most myeloma therapies for newly diagnosed patients.

DETAILED DESCRIPTION:
Induction Phase:

Newly diagnosed multiple myeloma patients with active disease, will be treated with Dd-R as outlined below:

All patients will also receive Levaquin 500 mg by mouth (PO) every day (QD) [or if allergic receive amoxicillin 250 mg PO twice a day (BID)], acyclovir 400 mg PO BID or Valacyclovir 500 mg BID and aspirin 81 mg PO QD daily while receiving Dd-R. Aspirin will continue through maintenance. For patients who cannot tolerate aspirin, low molecular weight heparin or therapeutic doses of coumadin may be used in place of aspirin.

* Doxil® 30 mg/m^2 on day # 1 to be repeated every 28 days
* Dexamethasone 40 mg per day for 4 days (days 1-4) every 28 days
* Revlimid® 25 mg PO daily on days 1-21, followed by 7 days of no therapy, repeated every 28 days

Maintenance Therapy:

Patients who complete the induction regimen or those who complete at least 2 cycles of the induction regimen and not showing evidence of progressive disease but cannot tolerate any further chemotherapy could be started on maintenance therapy as follows:

* Revlimid® 15 mg or 25 mg* PO daily on days 1-21, followed by 7 days of no therapy, repeated every 28 days

Patients will start maintenance therapy at the dexamethasone dose that was tolerated at the completion of the induction phase. *The starting Revlimid® dose for maintenance will be either 15 mg or 25 mg, which will be determined based on whether specific criteria are met on scheduled Day 1.

* Dexamethasone 40 mg per day for 4 days (days 1-4) every 28 days

All participants will also receive aspirin 81 mg PO QD daily while receiving maintenance. For patients who cannot tolerate aspirin, low molecular weight heparin or therapeutic doses of coumadin may be used in place of aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Diagnosed with active multiple myeloma and be considered to have active disease
* Measurable myeloma paraprotein levels in serum (≥ 0.5 g/dL) or urine (≥ 0.2 g excreted in a 24-hour urine collection sample).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Performance status of 3 will be allowed if related to bony disease.
* Prior steroid therapy for up to 4 weeks will not exclude the patient from entering the study.
* Bilirubin < 3.0
* Liver enzymes: alanine transaminase or aspartate transaminase (ALT or AST) < 3 x upper limit of normal (ULN)
* Must have adequate bone marrow function:
* Absolute neutrophil count > 1,000 cells/mm³ (1.0 x 10^9/L). Patients with bone marrow >50% plasma cells are permitted to have a neutrophil count of < 1,000 cells/mm³.
* Platelets ≥ 50,000 cells/mm³. Patients with bone marrow >50% plasma cells are permitted to have a Platelet count < 50, 000 cells/mm³.
* Hemoglobin > 8 g/dL (transfusion allowed to increase the Hgb)
* Must have adequate renal function: Creatinine ≤ 2.5 mg/dL
* Must have a 2-d echocardiogram indicating left ventricular ejection fraction (LVEF) ≥ 50% within 42 days prior to first dose of study drug
* Able to tolerate aspirin, low molecular weight heparin or coumadin
* Must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control AT THE SAME TIME, at least 4 weeks before taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy.

Exclusion Criteria:

* Ongoing severe infection requiring intravenous antibiotic treatment
* Life expectancy of <3 months
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the subject has been disease-free for at least 5 years. Concurrent prostate cancer for which the patient is receiving therapy will not be considered an exclusion if the prostatic specific antigen (PSA) has been stable for three years.
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
* Patients receiving therapeutic dosages of steroids (dexamethasone 160mg per pulse > 4 pulses) for multiple myeloma.
* Myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
* Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias), pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Prior chemotherapy for multiple myeloma, except for radiation to symptomatic bony disease, plasmapheresis for hyperviscosity, kyphoplasty and/or vertebroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachid Baz, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Baz RC, Shain KH, Hussein MA, Lee JH, Sullivan DM, Oliver EF, Nardelli LA, Nodzon LA, Zhao X, Ochoa-Bayona JL, Nishihori T, Dalton WS, Alsina M. Phase II study of pegylated liposomal doxorubicin, low-dose dexamethasone, and lenalidomide in patients with newly diagnosed multiple myeloma. Am J Hematol. 2014 Jan;89(1):62-7. doi: 10.1002/ajh.23587. PMID 24030918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 Eligible participants were enrolled at Moffitt Cancer Center between February 2008 and February 2011.
Period: Overall Study
Arm/Group | Induction and Maintenance Therapy
Started | 57
Completed | 47
Not Completed | 10
Not completed — Withdrew consent during Induction | 4
Not completed — Withdrew consent during Maintenance | 6

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Induction and Maintenance Therapy: Induction Phase Followed by Maintenance Therapy.
  Patients received lenalidomide 25 mg orally on days 1-21, dexamethasone 40 mg orally on days on 1-4, and PLD 40 mg/m^2 intravenously on day 1 (reduced to 30 mg/m^2 after the initial 29 patients were treated). Cycles were repeated every 28 days.
  At the best response (4-8 cycles of induction), patients could proceed with either high-dose therapy or maintenance with lenalidomide and dexamethasone at the tolerated doses on the same schedule until disease progression.
  Dd-R: Lenalidomide (Revlimid®) combined with Pegylated Liposomal Doxorubicin (Doxil®) and Dexamethasone (Decadron®) as outlined in the Detailed Description.
Arm/Group | Induction and Maintenance Therapy
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 63 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) - Percentage of Participants With Partial Response or Better With Induction Regimen
Description: ORR assessed using International Myeloma Working Group Response Definitions. Partial Remission (PR): A greater than 50% reduction in the serum paraprotein, and if present, a greater than 90% reduction in the urine M protein excretion. Patients must also have a decrease by 50% in the size of soft tissue plasmacytoma. If serum and urine M protein are not measurable, a 50% or greater decreased in the difference of the involved and uninvolved free light chain. Very Good Partial Remission (VGPR): Detectable serum and urine M component on immunofixation but not on electrophoresis or 90% or greater reduction in serum M protein with less than 100 mg/24 h of urinary M protein. Complete Remission (CR): The presence of less than 5% bone marrow plasmacytosis and the disappearance of all evidence of serum and urine M-components on electrophoresis as well as by immunofixation. In addition, soft tissue plasmacytoma must have disappeared.
Time Frame: 24 Months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Induction and Maintenance Therapy
Number analyzed (Participants) | 57
percentage of participants | 77.2

2. Primary Outcome: Percentage of Participants With Very Good Partial Remission (VGPR) or Better
Description: Quality of response: % Complete Response (CR) + Very Good Partial Remission (VGPR) to induction Dd-R as assessed using International Myeloma Working Group Response Definitions. Very Good Partial Remission (VGPR): Detectable serum and urine M component on immunofixation but not on electrophoresis or 90% or greater reduction in serum M protein with less than 100 mg/24 h of urinary M protein. Complete Remission (CR): The presence of less than 5% bone marrow plasmacytosis and the disappearance of all evidence of serum and urine M-components on electrophoresis as well as by immunofixation. In addition, soft tissue plasmacytoma must have disappeared.
Time Frame: 24 Months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Induction and Maintenance Therapy
Number analyzed (Participants) | 57
percentage of participants | 42.1

3. Secondary Outcome: Median Progression Free Survival (PFS) in Months
Description: PFS: Time from study entry to progression/relapse or death from study entry to death of any cause, assessed using International Myeloma Working Group Response Definitions. Progressive Disease (PD): One of the following criteria must be met: a. Increase of 25% or greater in serum M protein (absolute increase greater or equal to 0.5g/dl); b. Increase of 25% or greater in urine M protein (absolute increase greater than 200 mg/24h); c. Increase of 25% or greater in the difference between the involved and uninvolved free light chain (absolute increase greater than 10 mg/dl); d. Increase of 25% or greater in bone marrow plasma cell percentage (absolute percent greater than 5% in case the patient was in CR and 10% otherwise); i.e. Definite development of new bone lesions or soft tissue plasmacytomas, or increase in the size of existing plasmacytomas by greater or equal to 25%. Development of hypercalcemia (serum calcium > 11.5 mg/dl) attributable only to the plasma cell dyscrasia.
Time Frame: 24 Months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Maintenance Therapy
Number analyzed (Participants) | 57
months | 28 [18.1 to 34.8]

4. Secondary Outcome: 2 Year Overall Survival (OS) Rate
Description: Percentage of participants with Overall Survival in response to Dd-R in newly diagnosed multiple myeloma patients with active disease. Overall survival is time from study entry to death of any cause.
Time Frame: 24 Months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Induction and Maintenance Therapy
Number analyzed (Participants) | 57
percentage of participants | 79.6

5. Secondary Outcome: Occurrence of Induction Toxicities
Description: Tolerability of full dose Revlimid® with full dose Doxil® in combination with reduced schedule dexamethasone was to be assessed during Cycle 1 and at the start of Cycle 2 using, whenever possible, the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) v3.0.
  Due to increased neutropenia and fatigue, toxicities were reviewed after the first 29 participants were enrolled.
Time Frame: 24 Months
Population: First 29 participants with the PLD starting dose of PLD 40 mg/m^2, due to increased neutropenia and fatigue.
Measure: Number; unit: percentage of participants
Groups:
- Induction at Initial Full Dose: Induction Phase for First 29 Participants
  Patients received lenalidomide 25 mg orally on days 1-21, dexamethasone 40 mg orally on days on 1-4, and Pegylated Liposomal Doxorubicin (PLD) 40 mg/m^2 intravenously on day 1.
Arm/Group | Induction at Initial Full Dose
Number analyzed (Participants) | 29
percentage of participants
  Percentage with Dose Reductions Required | 24
  Percentage Receiving < 4 Cycles of Therapy | 20
  Percentage Who Discontinued After Only 1 Cycle | 13.79
  Percentage with Grade 3/4 Neutropenia | 48
  Percentage with Grade 3/4 Fatigue | 20

ADVERSE EVENTS:
Time Frame: 4 years, 10 months
Arm/Group | Induction and Maintenance Therapy
Serious Adverse Events (participants affected / at risk) | 26/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Maintenance Therapy (N=57)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Atrial (Cardiac disorders) | 1 (1)
Cardiac General - Other (Cardiac disorders) | 2 (2)
Constitutional Symptoms - Other (General disorders) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L) (General disorders) | 4 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 2 (2)
Infection(documented clinically or microbiologically) w/Grade 3 or 4 neutrophils - Lung(pneumonia) (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Sinus (Infections and infestations) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Foreign body (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Pain - NOS (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Syndromes - Other (General disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Maintenance Therapy (N=57)
Fatigue (General disorders) | 35 (60)
Sweating (diaphoresis) (General disorders) | 17 (17)
Fever (in the absence of neutropenia) (General disorders) | 13 (15)
Insomnia (General disorders) | 14 (16)
Rigors/chills (General disorders) | 12 (14)
Weight Loss (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 25 (35)
Diarrhea (Gastrointestinal disorders) | 24 (32)
Nausea (Gastrointestinal disorders) | 23 (33)
Anorexia (Gastrointestinal disorders) | 17 (20)
Gastrointestinal - Other (Gastrointestinal disorders) | 8 (15)
Vomiting (Gastrointestinal disorders) | 12 (17)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 12 (16)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 7 (7)
Heartburn/dyspepsia (Gastrointestinal disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 5 (6)
Dry mouth/salivary gland (Gastrointestinal disorders) | 4 (4)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5 (5)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 42 (238)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 41 (244)
Hemoglobin (Blood and lymphatic system disorders) | 25 (82)
Platelets (Blood and lymphatic system disorders) | 26 (111)
Lymphopenia (Blood and lymphatic system disorders) | 5 (20)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 21 (30)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 9 (14)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 5 (5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 8 (10)
Flushing (Skin and subcutaneous tissue disorders) | 5 (10)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (6)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pain - Head/headache (General disorders) | 11 (11)
Pain - Extremity-limb (General disorders) | 5 (6)
Pain - Abdomen NOS (General disorders) | 5 (5)
Pain - Throat/pharynx/larynx (General disorders) | 4 (6)
Pain - Joint (General disorders) | 3 (5)
Pain - Muscle (General disorders) | 3 (3)
Pain - Oral cavity (General disorders) | 4 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dizziness (General disorders) | 12 (12)
Neuropathy: sensory (Nervous system disorders) | 13 (16)
Mood alteration - Depression (Psychiatric disorders) | 7 (7)
Neurology - Other (Nervous system disorders) | 6 (6)
Syncope (fainting) (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 7 (7)
Neuropathy: motor (Nervous system disorders) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 29 (44)
Lymphatics - Other (Blood and lymphatic system disorders) | 3 (5)
Edema: head and neck (Blood and lymphatic system disorders) | 3 (4)
Febrile neutropenia (Infections and infestations) | 8 (11)
Infection with normal ANC or Grade 1 or 2 neutrophils - Vagina (Infections and infestations) | 3 (3)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 10 (16)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 9 (10)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 3 (3)
Allergic rhinitis (Immune system disorders) | 8 (8)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (8)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (10)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3 (3)
Hypotension (Cardiac disorders) | 7 (11)
Ocular/Visual - Other (Eye disorders) | 5 (5)
Dry eye syndrome (Eye disorders) | 3 (3)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Flu-like syndrome (General disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes